# ClinicalTrials.gov PRS DRAFT Receipt (Working Version) Last Update: 03/18/2021 14:27

#### ClinicalTrials.gov ID: NCT04184336

#### Study Identification

Unique Protocol ID: MENING

Brief Title: Enhanced Population-based Core Surveillance of Meningococcal Invasive

Infections at Participating Centers Across Canada

Official Title: IMPACT Project Protocol: Enhanced Population-based Core Surveillance of

Meningococcal Invasive Infections at Participating Centers Across Canada

Secondary IDs:

## **Study Status**

Record Verification: March 2021

Overall Status: Recruiting

Study Start: January 2016 [Actual]

Primary Completion: December 31, 2022 [Anticipated]

Study Completion: December 31, 2022 [Anticipated]

#### Sponsor/Collaborators

Sponsor: Canadian Paediatric Society

Responsible Party: Sponsor

Collaborators: Pfizer

### Oversight

U.S. FDA-regulated Drug: No

U.S. FDA-regulated Device: No

U.S. FDA IND/IDE: No

Human Subjects Review: Board Status: Approved

Approval Number: 1002978

Board Name: Research Ethics Board

Board Affiliation: IWK Health Center research services

Phone: 1-902-470-7879

Email: Address:

Data Monitoring: No